CLINICAL TRIAL: NCT04001868
Title: Immediate Effect of Sub Occipital Inhibition Technique on Postural Balance: Stabilometric Study.
Brief Title: Sub Occipital Inhibition Technique on Postural Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU UCH 212
Record Dates: First submitted 2019-06-19; First posted 2019-06-28 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Simple blind with evaluator blinded strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Application of the sub occipital inhibition technique.
  Interventions: Procedure: Suboccipital inhibition
- Placebo Group (Placebo Comparator): Hand contact in the sub occipital region without executing any technique.
  Interventions: Procedure: Placebo technique

INTERVENTIONS:
Procedure: Suboccipital inhibition — With the patient in the supine position and the therapist sitting at the head of the bed with the elbows resting on its surface. The therapist palpates the cervical spinous processes and slides the fingers upwards until contacting the posterior projection of the posterior arch of the atlas. Then, flexing the metacarpophalangeal at 90 degrees slowly raises the skull. The therapist's hands should remain together and the base of the skull should rest on his palms pressing with the index, middle and ring fingers of each hand in a sustained manner, but without causing pain. This pressure must be maintained during 4 minutes.
  Arms: Experimental Group
Procedure: Placebo technique — A superficial contact in the same area as the intervention, to rule out the exteroceptive effect associated with the therapist's contact.
  Arms: Placebo Group

SUMMARY:
In the present study the investigators want to verify if the inhibition of the suboccipital muscles improves the postural balance in subjects with cervical pain objectified by stabilometry.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who suffer neck pain for at least 3 months
* Come to receive physiotherapy treatment at Clinica Osteomed (NRS: 8415-CV), Elche, Alicante, Spain.
* Age between 18 and 65 years old.
* Sign the informed consent.

Exclusion Criteria:

* Suffering or having suffered pathologies of the postural control system (postural sensors, central nervous system or locomotor system)
* Presenting deformities or orthopedic injuries in the lower limbs or rachis
* Presenting pain at the moment of study
* Present contraindications to the intervention under study
* Have received physiotherapy treatment in the last six months
* Have undergone surgical treatment of any kind.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Surface of the ellipse open eyes | Postintervention immediate
  Determines the surface of the ellipse formed from the oscillations in the X and Y coordinates with open eyes. The measurement is made using a stabilometric platform with 4 pressure sensors per square centimeter. The software of the stabilometric platform collects 40 measurements per second through its pressure sensors, calculating the position of the projection of the center of gravity on the ground 40 times every second. The described variable evaluates the surface of the ellipse that contains the successive points of the displacement of the projection of the center of gravity in the ground during the standarized time for the stabilometric recording (51.2 seconds). It is a unique value, measured in a single moment. If the ellipse formed is larger, it implies a greater amplitude of the displacement of the center of gravity, and therefore a lower equilibrium capacity. Interval: 0-1000 (mm2).
Surface of the ellipse closed eyes | Postintervention immediate
  Determines the surface of the ellipse formed from the oscillations in the X and Y coordinates with closed eyes. The measurement is made using a stabilometric platform with 4 pressure sensors per square centimeter. The software of the stabilometric platform collects 40 measurements per second through its pressure sensors, calculating the position of the projection of the center of gravity on the ground 40 times every second. The described variable evaluates the surface of the ellipse that contains the successive points of the displacement of the projection of the center of gravity in the ground during the standarized time for the stabilometric recording (51.2 seconds). It is a unique value, measured in a single moment. If the ellipse formed is larger, it implies a greater amplitude of the displacement of the center of gravity, and therefore a lower equilibrium capacity. Interval: 0-1000 (mm2).

SECONDARY OUTCOMES:
Mean of the oscillation on the X axis and on the Y axis. | Preintervention and Postintervention immediate.
  It assesses the lateral and anteroposterior oscillation of the projection on the floor of the center of gravity during the 51 seconds of the stabilometric record. Interval: 0-50 (mm). Greater oscillation implies less postural balance.
Speed of the oscillation on the X axis and on the Y axis | Preintervention and Postintervention immediate.
  Determines the speed with which the projection of the center of gravity moves in lateral and anteroposterior direction during the 51 seconds of the stabilometric record. Interval: 0-10 (mm/s). Greater speed implies less postural balance.
Average speed of the oscillation | Preintervention and Postintervention immediate.
  Determines the average speed with which the projection of the center of gravity moves in lateral and anteroposterior direction during the 51 seconds of the stabilometric record. Interval: 0-10 (mm/s). Greater speed implies less postural balance.
Length of oscillation | Preintervention and Postintervention immediate.
  Determine the length of movement described by the projection on the ground of the center of gravity during the stabilometric measurement. Interval: 0-1000 (mm). Greater length implies less postural balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceu Cardenal Herrera University, Moncada, Valencia, Spain

REFERENCES:
- See also: The University CEU Cardenal Herrera is the first private university in the Valencia Community. It belongs to the Foundation San Pablo - CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04001868/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04001868/ICF_001.pdf